CLINICAL TRIAL: NCT07007676
Title: Effect of contINuous Glucose moniToring System on glycEmic controL in Non-insuLin-Treated Elderly People With Type 2 Diabetes: a Randomized Controlled Trial
Brief Title: Effect of Continuous Glucose Monitoring System on Glycemic Control in Non-insulin-Treated Elderly People With Type 2 Diabetes
Acronym: INTELLECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 6th People's Hospital (Other)
Collaborators: Shenzhen Center for Chronic Disease Control (Other); Shenzhen Baoan District People 's Hospital (Unknown); Shenzhen Haile Community Health Service Station (Unknown); Shenzhen Buxin Community Health Service Center (Unknown); Shenzhen Dalang Community Health Service Center (Unknown); Shenzhen Haihua Community Health Service Center (Unknown); Shenzhen Pingzhou Community Health Service Center (Unknown)
Responsible Party: Principal Investigator, Jian Zhou, Professor, Chief Physician, Deputy Director, Shanghai 6th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20250522001
Record Dates: First submitted 2025-05-23; First posted 2025-06-06 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus Type 2
Keywords: continuous glucose monitoring; non-insulin-treated; type 2 diabetes in the elderly
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real-time Continuous Glucose Monitoring （CGM） group (Experimental): CGM group participants will be asked to use a CGM sensor every 2 months. Participants will be instructed to use the sensor. In addition, participants will be advised to check the blood glucose when symptoms or expectations do not match the CGM reading.
  Interventions: Device: real-time CGM
- Blood Glucose Meter （BGM） group (No Intervention): BGM group participants will be asked to use a study blood glucose meter with test strips for a fingerstick blood glucose check with a recommendation of 2 times a week. Participants will be permitted to check a fingerstick glucose as many times a week as they choose.

INTERVENTIONS:
Device: real-time CGM — real-time CGM can provide real-time tracking of glucose levels, and offer glucose trend graphs and user-configurable low and high glucose alerts.
  Other Names: rtCGM; RT-CGM
  Arms: Real-time Continuous Glucose Monitoring （CGM） group

SUMMARY:
The goal of this clinical trial is to learn if continuous glucose monitoring system works to improve glucose control in non-insulin-treated older adults with type 2 diabetes. The main questions it aims to answer are:

* Dose the use of continuous glucose monitoring system improve glucose control in older adults with type 2 diabetes treated with oral antidiabetic drugs only?
* Dose the use of continuous glucose monitoring system affect psychological outcomes in older adults with type 2 diabetes treated with oral antidiabetic drugs only? Researchers will compare continuous glucose monitoring to standard blood glucose monitoring to see if continuous glucose monitoring works better in glucose management.

Participants will:

* Wear continuous glucose monitoring every 2 months or standard blood glucose monitoring for 6 months
* Visit the clinic once every 2 months for follow-up
* Keep a diary of their blood glucose when continuous glucose monitoring was not used

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years at the time of screening;
* Diagnosed with type 2 diabetes mellitus;
* Treated with two or more oral antidiabetic drugs with a stable medication regimen (medication classes) during the 3 months prior to entry;
* Suboptimal glycemic control, defined as HbA1c ≥ 7.5% and ≤ 10% at screening or within 30 days prior to screening visit;
* Has a smart phone compatible with CGM and BGM systems;
* Willing and able to provide written informed consent;
* At least 240 hours (10 out of 14 days) of sensor glucose data from the blinded CGM pre-randomization phase.

Exclusion Criteria:

* Use of insulin or Glucagon-Like Peptide-1 （GLP-1） receptor agonists within 3 months prior to screening;
* Use of any CGM device within 3 months prior to screening;
* Participants were unable to tolerate tape adhesive around sensor placement area, or with medically documented allergy towards the adhesive (glue) of plasters, or with serious skin diseases (e.g. psoriasis vulgaris, bacterial skin diseases) around sensor placement area;
* Considered unsuitable for participation by the investigators, including but not limited to individuals with dementia, psychiatric disorders, extreme visual or hearing impairment that would impair ability to use real-time CGM assessed;
* Planned surgery or other procedures within the next 6 months that may interfere with scheduled follow-up visits;
* Current or anticipated acute uses of glucocorticoids (oral, injectable, or IV), that will affect glycemic control;
* Estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73m2;
* Participation in any other clinical trial within 3 month prior to screening, or concurrently enrolled, or planning to participate in another trial during the study period.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | 24 weeks from baseline
  Change in HbA1c from baseline to 24 weeks

SECONDARY OUTCOMES:
Time in range of 70-180 mg/dL | 24 weeks from baseline
  A treatment group comparison of percentage of time spent in glucose range between 70 and 180 mg/dL measured by CGM
Time below range of 70 mg/dL | 24 weeks from baseline
  A treatment group comparison of percentage of time spent in glucose range below 70 mg/dL measured by CGM
Time above range of 180 mg/dL | 24 weeks from baseline
  A treatment group comparison of percentage of time spent in glucose range above 180 mg/dL measured by CGM
Glucose coefficient of variability | 24 weeks from baseline
  A treatment group comparison of glucose coefficient of variability measured by CGM
Mean glucose | 24 weeks from baseline
  A treatment group comparison of the mean glucose measured by CGM

OTHER OUTCOMES:
HbA1c <7.0% | 24 weeks from baseline
  Percentage of subjects with A1C less than 7%
Reduction in HbA1c ≥0.5% | 24 weeks from baseline
  Percentage of subjects with a reduction in A1C greater than or equal to 0.5%
Rate of hypoglycemia events per week | 24 weeks from baseline
  Hypoglycemia event was defined as 15 consecutive minutes with a sensor glucose value <70 mg/dL
Time in tight range of 70-140 mg/dL | 24 weeks from baseline
  A treatment group comparison of the percentage of time spent in glucose range between 70 and 140 mg/dL measured by CGM
Glycemia risk index (GRI) | 24 weeks from baseline
  A treatment group comparison of the glycemia risk index measured by CGM. Glycemia risk index (GRI) was calculated according to the following equation: GRI = (3.0×VLow) + (2.4×Low) + (1.6×VHigh) + (0.8×High).
Glucose standard deviation | 24 weeks from baseline
  A treatment group comparison of the glucose standard deviation measured by CGM
Days to initiate inulin treatment | 24 weeks from baseline
  A treatment group comparison of the days to initiate inulin treatment during study period
Change in the scores of psychological-related questionnaires | 24 weeks from baseline
  Psychological-related events were measured by Diabetes Distress Scale and Patient Health Questionnaire-8 items.
Change in the score of blood glucose monitoring satisfaction questionnaire | 24 weeks from baseline
  Change in the score of blood glucose monitoring satisfaction questionnaire from 24 weeks from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, Prof., Dr., Ph.D, Principal Investigator — Shanghai 6th People's Hospital; Xiaobing Wu, Ph.D, Principal Investigator — Shenzhen Center for Chronic Disease Control
Locations (5):
- China (5):
  - Shenzhen Buxin Community Health Service Center, Shenzhen, Guangdong
  - Shenzhen Dalang Community Health Service Center, Shenzhen, Guangdong
  - Shenzhen Haihua Community Health Service Center, Shenzhen, Guangdong
  - Shenzhen Haile Community Health Service Station, Shenzhen, Guangdong
  - Shenzhen Pingzhou Community Health Service Center, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: No